CLINICAL TRIAL: NCT07206719
Title: Safety and Efficacy of Concurrent MACE and Mitrofanoff Procedures for Management of Neuropathic Fecal and Urinary Incontinence in Children
Brief Title: Safety and Efficacy of Concurrent MACE and Mitrofanoff Procedures
Acronym: MitroMACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammad Daboos (Other)
Responsible Party: Sponsor-Investigator, Mohammad Daboos, Assistant professor of pediatric surgery, Pediatric Surgery Department, Al-Azhar University., Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 67-Med-0000072-8-01-022; 0000072-8-01-022 (Other: Al Azhar University)
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Fecal Incontinence; Urinary Incontinence
Keywords: Urinary incontinence; Fecal incontinence; Quality of life; Mitrofanoff procedure; Malone procedure
MeSH Terms: conditions — Fecal Incontinence; Urinary Incontinence | interventions — omega-Chloroacetophenone

STUDY DESIGN:
Intervention Model Description: MACE Split appendix procedure:
  MACE Colonic flap Neoappendecosotomy procedure
  Mitrofanoff procedure:
Masking Description: surgical management by concurrent Malone Antigrade Continent Enema (MACE) and Mitrofanoff procedures at the same operative sitting, for patients suffered from combined fecal and urinary incontinence due to neuropathic etiology.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MACE and Malone (Experimental): patients suffering from combined fecal and urinary incontinence due to neuropathic etiology, after failure of all trials of non-surgical managements. They submitted for surgical management by concurrent Malone Antegrade Continent Enema (MACE) and Mitrofanoff procedures at the same operative sitting
  Interventions: Procedure: Malone Antegrade Continent Enema (MACE) and Mitrofanoff procedures

INTERVENTIONS:
Procedure: Malone Antegrade Continent Enema (MACE) and Mitrofanoff procedures — * MACE Split appendix procedure: division of appendix into two segments, so making Mitrofanoff procedure by the distal appendicular segment and Malone procedure by proximal appendicular segment.
  * MACE Colonic flap Neoappendecosotomy procedure: creating the colonic flap from the ascending colon, tubularization done. The tip of the neo-appendix was spatulated and sutured with the triangular skin flap of umbilicus, then the silicon catheter in place passing through the neo appendix into the colon
  * Mitrofanoff procedure: The appendix was mobilized with its mesentery. The tip of the appendix was incised and a 10-12Fr feeding tube was inserted to confirm patency. Then Opening of the urinary bladder was done. The distal end of the appendix was then inserted into the bladder in a submucosal tunnel. The distal opening of the appendix was sutured to the inner bladder wall and mucosa using absorbable sutures.

SUMMARY:
This was a prospective study. The study period was from January 2022 to July 2025. The study included 30 patients suffering from combined fecal and urinary incontinence submitted for concurrent Malone Antigrade continent Enema and Mitrofanoff procedures and evaluated regarding intraoperative difficulties, post-operative complications, functional results and patient's quality of live improvements.

DETAILED DESCRIPTION:
-This was a prospective study, at Al-Azhar university hospitals. The study period was from January 2022 to July 2025. The study included all patients suffering from combined fecal and urinary incontinence after failure of all trials of non-surgical managements.

The investigator aimed to study the safety and surgical oucomes of the management of fecal and urinary incontinence in children by concurrent Malone Antigrade Continent Enema and Mitrofanoff procedures regarding intraoperative difficulties, post-operative complications, functional results and patient's quality of live improvements.

* They submitted for surgical management by concurrent Malone Antigrade Continent Enema (MACE) and Mitrofanoff procedures at the same operative sitting.
* the outcomes measures included:--Intraoperative parameters including length of appendix, operative time, and intraoperative complications (bleeding, visceral injury, ureteric injury, appendicular vascular affection).
* Postoperative parameters

  1. Early as Occurrence of leak, abscess formation, intestinal obstruction, appendicular necrosis, fecal and urinary fistula formation.
  2. Late as Stricture formation and requirement of secondary procedures as dribbling of urine through the urethra or soiling of stool. Also function result as volume of required colonic washout fluid, frequency of the Malone stoma catheterization, Frequency of Mitrofanoff catheterization, urine volume and Patient quality of life utilizing QOL score 9
* We started Mitrofanoff stoma catheterization after three weeks of procedure. and Started Malone ante grade continent enema after one month. The volume of saline used for washout was calculated according to body weight 20ml/kg. Outpatient clinic visits every week then at 3, 6 and 12 months postoperatively for evaluation of post-operative complications, function outcome and patient QOL score

ELIGIBILITY:
Inclusion Criteria:

* all patients suffering from combined fecal and urinary incontinence due to neuropathic etiology
* failure of all trials of non-surgical managements

Exclusion Criteria:

* The patients responding to medical treatments,
* patients with previous appendectomy,
* patients with marked reduction of bladder capacity,
* patients with Brain affection (Cerebral palsy, etc..)
* and patients with isolated fecal or urinary incontinence

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Surgical Outcomes | 6 months
  Complication rate
  1-Early as Occurrence of leak, abscess formation, intestinal obstruction, appendicular necrosis, fecal and urinary fistula formation.
  2. Late as Stricture formation and requirement of secondary procedures as dribbling of urine through the urethra or soiling of stool

SECONDARY OUTCOMES:
Patients Quality Of Life post operatively | 6 months
  Quality Of Life Score
  1. How would you describe your child's social habits?
  2. How would you describe your child's school attendance?
  3. How would you describe your child's daily activity?
  4. How would you describe your child's physical activity?
  5. Does your child spend the night in places other than your home?
  6. How would you describe how your child feels?
  7. How would you describe your child's relationships with peers (like classmates)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Daboos, prof, Principal Investigator — Al-Azhar University
Locations (1):
- Mohammad Daboos, Cairo, Egypt